CLINICAL TRIAL: NCT00497003
Title: Effect of Beta Blocker Treatment on Endothelial Function in Patients With Type 2 Diabetes or Chronic Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Danish Heart Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KF 02-071/03
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2007-10-15 (Estimated); Status verified 2007-07

CONDITIONS: Endothelial Function; Beta Blocker
Keywords: Endothelial function; Beta blocker; Type 2 diabetes; Chronic heart failure
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Therapeutics; Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Treatment with either metoprolol or carvedilol

SUMMARY:
The aim of this study is to evaluate the effect of the two different beta blockers metoprolol and carvedilol on endothelial function in patients with either type two diabetes or chronic heart failure.

Hypothesis: 1* Carvedilol compared to metoprolol has a favourable effect on endothelial function.

2* Carvedilol compared to metoprolol has a favourable effect on insulin stimulated endothelial function.

The study is conducted as an open parallel group study. Endothelial function and insulin stimulated endothelial function was evaluated before and after a two months treatment period with either of the two beta blockers.

DETAILED DESCRIPTION:
Endothelial function is deteriorated in patients with type 2 diabetes and in patients with chronic heart failure. Treatment with carvedilol improves survival in patients with chronic heart failure compared to treatment with metoprolol. Carvedilol improves metabolic glucose control in patients with diabetes compared to metoprolol.Carvedilol compared to metoprolol also decreases the number of patients with new onset diabetes among patients with chronic heart failure. The mechanism behind these findings has not been fully understood.

The purpose of this study is to investigate if carvedilol compared to metoprolol has a favourable effect on endothelial function and insulin stimulated endothelial function, in groups of patients with either diabetes or chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Chronic heart failure

Exclusion Criteria:

* For patients with type 2 diabetes:

  * Vascular complications.
* For patients with chronic heart failure:

  * Severe uncontrolled heart failure.
  * Untreated severe hypertension, hypotension.
  * Bradycardia.
  * Known intolerance to beta blocker treatment.
  * Pregnancy,

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-02; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Endothelial function and insulin stimulated endothelial function | 2 months

SECONDARY OUTCOMES:
Insulin stimulated glucose uptake | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Torp-Pedersen, MD, DSc, Principal Investigator — Department of Cardiology, Bispebjerg Hospital
Locations (1):
- Department of Cardiology, University Hospital of Copenhagen, Bispebjerg, Copenhagen, Denmark

REFERENCES:
- [Derived] Falskov B, Hermann TS, Raunso J, Christiansen B, Rask-Madsen C, Major-Pedersen A, Kober L, Torp-Pedersen C, Dominguez H. Endothelial function is unaffected by changing between carvedilol and metoprolol in patients with heart failure--a randomized study. Cardiovasc Diabetol. 2011 Oct 15;10:91. doi: 10.1186/1475-2840-10-91. PMID 21999413
- [Derived] Kveiborg B, Hermann TS, Major-Pedersen A, Christiansen B, Rask-Madsen C, Raunso J, Kober L, Torp-Pedersen C, Dominguez H. Metoprolol compared to carvedilol deteriorates insulin-stimulated endothelial function in patients with type 2 diabetes - a randomized study. Cardiovasc Diabetol. 2010 May 25;9:21. doi: 10.1186/1475-2840-9-21. PMID 20500877